CLINICAL TRIAL: NCT03536104
Title: Identification of Risk Factors Parkinson's Disease by Convergence Strategy
Acronym: CONVERGENCE
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2008_0811; 2008-A00219-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-05-14; First posted 2018-05-24 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, CSF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Controls: This group will include "healthy" person.
- Parkinson's patient: This group will include Parkinsonian patients
- patients with a related disease.: This group will include patients with a related disease.

SUMMARY:
Using this convergence approach from a limited group of subjects with non-diseased controls, patients with Parkinson's disease or related diseases, we will be able to limit the number of potential genes of specific susceptibility to Parkinson disease. These genes will then be studied using a case-control genetic epidemiology approach. The risk of developing the disease will then be evaluated according to clinical, biological and environmental variables collected in Parkinson's subjects and healthy controls in the second group of subjects. The specificity of the genetic associations found will be evaluated in subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for Parkinson's patients and "related diseases" controls:
* Parkinsonian patients meeting the Gelb criteria
* Patients with other neurodegenerative disease (such as other Parkinson syndrome or synucleopathies) meeting the criteria set out in Appendix 2 (Lewy Bodies dementia, Parkinson's disease with dementia, MultiSystem atrophy, Progressive Supranuclear Paralysis) , Amyotrophic Lateral Sclerosis, Restless Legs Syndrome, Alzheimer's Disease).
* Woman of childbearing age having an effective means of contraception.
* Informed consent signed by the subject or his legal representative.
* For demented subjects coming for consultation or day hospitalization with an accompanying person, signature of the legal representative.

Criteria for inclusion of non-ill controls:

* Absence of rest trembling, bradykinesia and stiffness
* MMSE (Mini Mental State Examination) greater than 25
* Woman of childbearing age having an effective means of contraception.
* subject having signed the informed consent.
* No family history of neurodegenerative disease that started before age 70. These controls will not present any Parkinsonian signs during the clinical evaluation. They may have functional disabilities whose cause is known and unrelated to a neurodegenerative disease with a cognitive function measurement greater than 25 in the MMSE test.

Exclusion Criteria:

* Criteria for non-inclusion of patients:
* Clinical criteria for exclusion of the diseases described
* Participation in another therapeutic trial or in the exclusion period of a previous clinical trial.

Criteria for non-inclusion of non-ill controls:

* Functional discomfort in daily life of unknown cause
* MMSE less than 25
* Participation in another therapeutic trial or in the exclusion period of a previous clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson Disease compared to subjects at risk to develop Parkinson Disease and healthy controls
Sampling Method: Probability Sample
Enrollment: 2220 (Actual)
Dates: Start 2009-03-25 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

PRIMARY OUTCOMES:
Significant variations in the frequencies of gene polymorphisms and the risk of developing Parkinson's disease | through study completion, an average of 10 years
  the frequency is measured according to biological and environmental variables modulating the risk of developing Parkinson's disease.

CONTACTS AND LOCATIONS:
Overall Officials: Alain DESTEE, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Roger Salengro, CHRU de Lille, Lille, France

IPD SHARING:
Plan to Share IPD: No